CLINICAL TRIAL: NCT01461811
Title: ARES Registration Trial
Brief Title: Prospective Study of an Investigational Toric Soft Contact Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CIBA VISION (Industry)
Responsible Party: Sponsor
Organization: Alcon Research (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: C-11-035 (P-415-C-003)
Record Dates: First submitted 2011-10-26; First posted 2011-10-28 (Estimated); Results first posted 2013-10-17 (Estimated); Last update posted 2013-10-17 (Estimated); Status verified 2013-08

CONDITIONS: Myopia; Astigmatism; Refractive Error
Keywords: toric; contact lenses; daily disposable contact lenses; astigmatism; soft contact lenses; contact lens comfort
MeSH Terms: conditions — Myopia; Astigmatism; Refractive Errors

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- DAILIES® AquaComfort Plus® Toric (Experimental): Nelfilcon A toric contact lenses (with comfort additives) worn in both eyes on a daily wear, daily disposable basis for three months
  Interventions: Device: Nelfilcon A toric contact lenses (with comfort additives)
- Focus® DAILIES® Toric (Active Comparator): Nelfilcon A toric contact lenses worn in both eyes on a daily wear, daily disposable basis for three months
  Interventions: Device: Nelfilcon A toric contact lenses

INTERVENTIONS:
Device: Nelfilcon A toric contact lenses (with comfort additives)
  Arms: DAILIES® AquaComfort Plus® Toric
Device: Nelfilcon A toric contact lenses
  Other Names: Focus® DAILIES® Toric
  Arms: Focus® DAILIES® Toric

SUMMARY:
The purpose of this study was to demonstrate substantial equivalence of an investigational toric soft contact lens to the commercially available Focus® DAILIES® Toric soft contact lens when worn in a daily wear, daily disposable mode for three months.

DETAILED DESCRIPTION:
Eligible participants were randomized 2:1 to wear either DAILIES® AquaComfort Plus® Toric or Focus® DAILIES® Toric.

ELIGIBILITY:
Inclusion Criteria:

* Sign Informed Consent document. If under legal age of consent, legally authorized representative must sign Informed Consent document and participant must sign Assent document.
* Normal eyes not using any ocular medications that would contraindicate lens wear.
* Willing and able to wear toric contact lenses in both eyes within the available range of powers for this trial.
* Spectacle cylinder prescription between 0.50 and 2.00 diopters.
* Best spectacle corrected visual acuity 20/25 (Snellen) or better in each eye at distance.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Anterior segment infection, inflammation, or abnormality.
* Any active anterior segment or systemic disease that would contraindicate contact lens wear.
* Use of systemic medications that would contraindicate lens wear.
* Any ocular or systemic medical condition that may, in the opinion of the investigator, preclude safe administration of the study lenses or affect the results of this study.
* History of herpetic keratitis.
* History of refractive surgery or irregular cornea.
* History of pathologically dry eye.
* Corneal vascularization greater than 1 mm of penetration.
* Eye injury within twelve weeks immediately prior to enrollment in this trial.
* Participation in a contact lens or contact lens care product clinical trial within the previous 30 days, or concurrent participation in any clinical trial.
* Other protocol-defined exclusion criteria may apply.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2011-12; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Fahmy, OD, Study Director — Alcon Research

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from ten US study centers.
Pre-assignment Details: Of the 154 participants enrolled, ten participants were considered enrolled, but not dispensed, due to not meeting inclusion criteria or withdrawal of consent. This reporting group includes all enrolled and dispensed participants (144).
Period: Overall Study
Arm/Group | DAILIES® AquaComfort Plus® Toric | Focus® DAILIES® Toric
Started | 95 | 49
Completed | 91 | 46
Not Completed | 4 | 3
Not completed — Adverse Event | 2 | 1
Not completed — Subject decision unrelated to an AE | 1 | 1
Not completed — Noncompliance | 1 | 1

BASELINE CHARACTERISTICS:
Population: This reporting group includes all enrolled and dispensed participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | DAILIES® AquaComfort Plus® Toric | Focus® DAILIES® Toric | Total
Number analyzed (Participants) | 95 | 49 | 144
Age Continuous [Mean (Standard Deviation); unit: years] | 33.6 (12.5) | 37.2 (11.4) | 34.9 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 73 | 28 | 101
  Male | 22 | 21 | 43

OUTCOME MEASURES:

1. Primary Outcome: Contact Lens-Corrected Distance Monocular Snellen Visual Acuity (VA) (20/30 or Better)
Description: Visual acuity, as assessed for each eye individually. Participant read a distance Snellen chart while wearing study lenses. The percentage of eyes with VA recorded as 20/30 or better is reported. Both eyes contributed to the percentage.
Time Frame: Up to Month 3
Population: All enrolled and dispensed participants, with exclusions due to reasons such as discontinuations and/or missing responses.
Measure: Number; unit: Percentage of eyes
Arm/Group | DAILIES® AquaComfort Plus® Toric | Focus® DAILIES® Toric
Number analyzed (Participants) | 91 | 46
Percentage of eyes
  Dispense | 98.9 | 98.9
  Week 1 | 98.9 | 97.8
  Week 2 | 98.9 | 97.8
  Month 1 | 98.9 | 97.8
  Month 2 | 98.9 | 98.9
  Month 3 | 98.9 | 96.7

2. Secondary Outcome: Subjective Rating of Insertion Comfort
Description: Insertion comfort (30 seconds to 1 minute), as rated by the participant on a 10-point scale, with 1 being poor and 10 being excellent. The participant rated both eyes together by providing one single rating.
Time Frame: Up to Month 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | DAILIES® AquaComfort Plus® Toric | Focus® DAILIES® Toric
Number analyzed (Participants) | 91 | 46
Units on a scale
  Dispense | 8.9 (1.3) | 9.0 (1.4)
  Week 1 | 9.0 (1.3) | 9.0 (1.4)
  Week 2 | 9.0 (1.1) | 9.1 (1.2)
  Month 1 | 9.0 (1.1) | 9.1 (1.1)
  Month 2 | 9.1 (0.9) | 9.3 (0.9)
  Month 3 | 9.2 (1.0) | 9.1 (1.3)

3. Secondary Outcome: Subjective Rating of End of Day Comfort
Description: End of day comfort, as rated by the participant on a 10-point scale, with 1 being poor and 10 being excellent. The participant rated both eyes together by providing one single rating.
Time Frame: Up to Month 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | DAILIES® AquaComfort Plus® Toric | Focus® DAILIES® Toric
Number analyzed (Participants) | 91 | 46
Units on a scale
  Week 1 | 7.2 (2.5) | 7.6 (2.1)
  Week 2 | 7.6 (2.1) | 7.9 (1.8)
  Month 1 | 7.6 (2.0) | 8.2 (1.4)
  Month 2 | 7.6 (2.1) | 7.9 (1.9)
  Month 3 | 7.7 (1.9) | 7.8 (2.0)

4. Secondary Outcome: Subjective Rating of Overall Comfort
Description: Overall comfort, as rated by the participant on a 10-point scale, with 1 being poor and 10 being excellent. The participant rated both eyes together by providing one single rating.
Time Frame: Up to Month 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | DAILIES® AquaComfort Plus® Toric | Focus® DAILIES® Toric
Number analyzed (Participants) | 91 | 46
Units on a scale
  Week 1 | 8.1 (1.7) | 8.7 (1.1)
  Week 2 | 8.3 (1.5) | 8.7 (1.3)
  Month 1 | 8.4 (1.4) | 8.8 (1.1)
  Month 2 | 8.2 (1.5) | 8.7 (1.2)
  Month 3 | 8.4 (1.4) | 8.7 (1.3)

5. Secondary Outcome: Subjective Rating of End of Day Dryness
Description: End of day dryness, as rated by the participant on a 10-point scale, with 1 being dry and 10 being not dry. The participant rated both eyes together by providing one single rating.
Time Frame: Up to Month 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | DAILIES® AquaComfort Plus® Toric | Focus® DAILIES® Toric
Number analyzed (Participants) | 91 | 46
Units on a scale
  Week 1 | 7.1 (2.7) | 7.1 (2.3)
  Week 2 | 7.2 (2.3) | 7.6 (2.1)
  Month 1 | 7.3 (2.0) | 7.9 (1.6)
  Month 2 | 7.4 (2.1) | 7.6 (2.0)
  Month 3 | 7.5 (2.0) | 7.4 (2.2)

6. Secondary Outcome: Subjective Rating of Overall Vision
Description: Overall vision, as rated by the participant on a 10-point scale, with 1 being poor and 10 being excellent. The participant rated both eyes together by providing one single rating.
Time Frame: Up to Month 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | DAILIES® AquaComfort Plus® Toric | Focus® DAILIES® Toric
Number analyzed (Participants) | 91 | 46
Units on a scale
  Dispense | 8.6 (1.4) | 8.9 (1.2)
  Week 1 | 8.7 (1.6) | 8.8 (1.1)
  Week 2 | 8.8 (1.4) | 8.9 (1.0)
  Month 1 | 8.7 (1.3) | 8.9 (0.9)
  Month 2 | 8.7 (1.4) | 8.9 (0.9)
  Month 3 | 8.9 (1.2) | 8.8 (1.3)

7. Secondary Outcome: Subjective Rating of Overall Handling
Description: Overall handling, as rated by the participant on a 10-point scale, with 1 being difficult and 10 being easy. The participant rated both eyes together by providing one single rating.
Time Frame: Up to Month 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | DAILIES® AquaComfort Plus® Toric | Focus® DAILIES® Toric
Number analyzed (Participants) | 91 | 46
Units on a scale
  Dispense | 9.0 (1.2) | 9.0 (1.7)
  Week 1 | 8.8 (1.4) | 8.7 (1.2)
  Week 2 | 9.0 (0.9) | 8.8 (1.2)
  Month 1 | 9.0 (1.2) | 8.9 (1.1)
  Month 2 | 9.0 (1.2) | 9.0 (1.1)
  Month 3 | 9.0 (1.1) | 9.1 (1.1)

8. Secondary Outcome: Lens Centration (Centered, Slight Decentration)
Description: Lens centration, as assessed by the investigator for each eye individually. Lens centration was graded on a 5-point scale: 0=centered, 1=slight decentration, 2=mild decentration, 3=moderate decentration, 4=severe decentration. The combined percentage of lenses assessed as "centered" or "slight decentration" is reported. Lenses from both eyes contributed to the percentage.
Time Frame: Up to Month 3
Population: as for outcome 1
Measure: Number; unit: Percentage of lenses
Arm/Group | DAILIES® AquaComfort Plus® Toric | Focus® DAILIES® Toric
Number analyzed (Participants) | 91 | 46
Percentage of lenses
  Dispense | 97.8 | 98.9
  Week 1 | 100 | 100
  Week 2 | 100 | 100
  Month 1 | 100 | 100
  Month 2 | 100 | 100
  Month 3 | 99.4 | 100

9. Secondary Outcome: Lens Fit (Optimal, Acceptably Loose, Acceptably Tight)
Description: Lens fit, as assessed by the investigator for each eye individually. Lens fit was graded on a 5-point scale: 2=unacceptably loose, 1=acceptably loose, 0=optimal, -1=acceptably tight, and -2=unacceptably tight. The combined percentage of lenses assessed as "optimal," "acceptably loose," or "acceptably tight" is reported. Lenses from both eyes contributed to the percentage.
Time Frame: Up to Month 3
Population: as for outcome 1
Measure: Number; unit: Percentage of lenses
Arm/Group | DAILIES® AquaComfort Plus® Toric | Focus® DAILIES® Toric
Number analyzed (Participants) | 91 | 46
Percentage of lenses
  Dispense | 100 | 100
  Week 1 | 100 | 100
  Week 2 | 100 | 100
  Month 1 | 100 | 100
  Month 2 | 100 | 100
  Month 3 | 100 | 100

10. Secondary Outcome: Front Surface Wettability (None, Very Slight)
Description: Front surface wettability (i.e., assessment of the disruption of the front surface wettability of the contact lens), as assessed by the investigator for each eye individually. Front surface wettability was graded on a 5-point scale: 0=none, 1=very slight, 2=slight, 3=moderate, 4=severe. The combined percentage of lenses assessed as "none" or "very slight" is reported. Lenses from both eyes contributed to the percentage.
Time Frame: Up to Month 3
Population: as for outcome 1
Measure: Number; unit: Percentage of lenses
Arm/Group | DAILIES® AquaComfort Plus® Toric | Focus® DAILIES® Toric
Number analyzed (Participants) | 91 | 46
Percentage of lenses
  Dispense | 99.4 | 100
  Week 1 | 92.2 | 97.8
  Week 2 | 94.9 | 95.6
  Month 1 | 97.2 | 93.5
  Month 2 | 91.1 | 86.7
  Month 3 | 91.6 | 88.0

11. Secondary Outcome: Front Surface Deposits (None, Very Slight)
Description: Front surface deposits on the contact lens, as assessed by the investigator for each eye individually. Front surface deposits were graded on a 5-point scale: 0=none, 1=very slight, 2=slight, 3=moderate, 4=severe. The combined percentage of lenses assessed as "none" or "very slight" is reported. Lenses from both eyes contributed to the percentage.
Time Frame: Up to Month 3
Population: as for outcome 1
Measure: Number; unit: Percentage of lenses
Arm/Group | DAILIES® AquaComfort Plus® Toric | Focus® DAILIES® Toric
Number analyzed (Participants) | 91 | 46
Percentage of lenses
  Dispense | 100 | 100
  Week 1 | 96.1 | 100
  Week 2 | 98.3 | 100
  Month 1 | 98.9 | 99
  Month 2 | 98.9 | 96.7
  Month 3 | 96.1 | 97.8

12. Secondary Outcome: Back Surface Debris/Deposits (None, Very Slight)
Description: Back surface debris/deposits on the contact lens, as assessed by the investigator for each eye individually. Back surface debris/deposits were graded on a 5-point scale: 0=none, 1=very slight, 2=slight, 3=moderate, 4=severe. The combined percentage of lenses assessed as "none" or "very slight" is reported. Lenses from both eyes contributed to the percentage.
Time Frame: Up to Month 3
Population: as for outcome 1
Measure: Number; unit: Percentage of lenses
Arm/Group | DAILIES® AquaComfort Plus® Toric | Focus® DAILIES® Toric
Number analyzed (Participants) | 91 | 46
Percentage of lenses
  Dispense | 100 | 100
  Week 1 | 98.9 | 100
  Week 2 | 100 | 100
  Month 1 | 100 | 100
  Month 2 | 96.6 | 96.7
  Month 3 | 99.4 | 98.9

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of consent and reported for the duration of the study.
Description: This reporting group includes all enrolled and dispensed participants.
Arm/Group | DAILIES® AquaComfort Plus® Toric | Focus® DAILIES® Toric
Serious Adverse Events (participants affected / at risk) | 0/95 | 0/49
Other Adverse Events (participants affected / at risk) | 0/95 | 0/49

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
For a period of 10 years, the clinical investigator must hold all trial-related information and documents confidential and must obtain sponsor's written consent before discussing, presenting, publicizing, or otherwise disclosing any preclinical and/or clinical data or impressions from this trial.